CLINICAL TRIAL: NCT04705584
Title: Role of Topical Immuonosuppressant in the Management of Spring Catarrh: a Comparative Study Between Cyclosporine A 2% and Tacrolimus 0.3%
Brief Title: Topical Immuonosuppressant Drugs in Spring Catarrh
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Zeiad Eldalyl, Lecturer of Ophthalmology, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17101246
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Vernal Keratoconjunctivitis
Keywords: Resistant spring catarrh; Cyclosporine A; Tacrolimus
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Topical steroids (Active Comparator): Topical Prednisolone acetate 1.0% Topical eye drops 4 times per day for 2 weeks followed by 4 times daily for 2 weeks, then twice daily for 2 weeks and finally once daily for 2 weeks.
  Interventions: Drug: Prednisolone (as Acetate)
- Topical Cyclosporine A (Experimental): Topical Prednisolone acetate 1.0% Topical eye drops 4 times per day for 2 weeks followed by Topical Cyclosporine A 2% Topical eye drops 2 times per day for 6 weeks.
  Interventions: Drug: CycloSPORINE Ophthalmic Suspension
- Topical Tacrolimus (Experimental): Topical Prednisolone acetate 1.0% Topical eye drops 4 times per day for 2 weeks followed by Topical Tacrolimus A 0.3% Topical eye drops 2 times per day for 6 weeks.
  Interventions: Drug: LTacrolimus Topical

INTERVENTIONS:
Drug: Prednisolone (as Acetate) — Standard treatment protocol includes Topical steroids for 8 weeks with gradual dose tapering.
  Other Names: Predforte Eye drops
  Arms: Topical steroids
Drug: CycloSPORINE Ophthalmic Suspension — This treatment arm includes the use of topical cyclosporine A after 2 weeks of topical steroid use.
  Arms: Topical Cyclosporine A
Drug: LTacrolimus Topical — This treatment arm includes the use of topical Tacrolimus after 2 weeks of topical steroid use.
  Arms: Topical Tacrolimus

SUMMARY:
Spring catarrh is a prevalent type of conjunctival allergic disorder in temperate countries. Topical steroids are the cornerstone management of spring catarrh beside other anti allergic drugs. However, prolonged use of topical steroids especqially in resistant spring catarrh carries risk of ocular side effects as 2nd glaucoma and cataract. We will investigate the safety and efficacy of topical immuonosuppressant in the management of resistant spring catarrh as an alternative to steroid therapy.

DETAILED DESCRIPTION:
Vernal keratoconjunctivitis (VKC) (spring catarrh) is an allergic disease that affects children and young adults and is one of the most severe forms of atopic ocular disease. Classically, the incidence of VKC peaks in the summer and spring. However, 60% of cases can become chronic with persistent symptoms. VKC is mainly characterized by intense itching, but patients also frequently complain of lacrimation, foreign body sensation and photophobia.

There are three different clinical forms of VKC; the palpebral form, which is characterized by giant papillae in the upper tarsal; the limbal form, with gelatinous nodules composed of eosinophilic infiltrates and degenerated epithelial cells (Horner- Tantra spots) and a mixed form.

The treatment of VKC involves the use of topical Anti-histaminic and Mast Cell Stabilizers, which are usually sufficient to control symptoms in mild cases. However, a high number of patients are refractory to allergy therapy and require treatment with topical steroids. Side effects related to long-term steroid use, such as increased intraocular pressure (IOP), cataract development and increased susceptibility to infections.

Refractory VKC, development of steroid complications or the need for long-term use of Topical steroids are indications to use Topical immune-suppressant drugs as Tacrolimus (TCL) or Cyclosporine A (CsA). Tacrolimus is an immunosuppressant derived from Streptomyces tsukubaensis, is an alternative to steroid therapy for allergic diseases of the ocular surface. Topical Cyclosporine A is a fungal metabolite that reduces ocular inflammation by inhibiting Th2 lymphocyte proliferation and histamine release from mast cells and basophils.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from Vernal Keratoconjunctivitis refractory to conventional treatments (Topical Anti-histaminic agents, Mast-cell stabilizer and steroids) are included.

Exclusion Criteria:

* Contact lens wearer. Patient with one functioning eye. Patients with any other active ocular inflammatory conditions. Patients with hypersentivity reaction to either Cyclosporine A or Tacrolimus. Loss of 2 or more follow up visits.

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-01 (Estimated); Primary Completion 2021-10 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Ocular surface changes | 8 weeks
  Changes in papillary conjunctival reaction, conjunctival redness, Tranta spots and gelatinous masses

SECONDARY OUTCOMES:
Ocular symptoms changes | 8 weeks
  Change of ocular symptoms as documented by the patient as redness, itching and discharge
Intraocular pressure changes | 8 weeks
  Mean change of intraocular pressure from baseline
Ocular surface toxicity | 8 weeks
  Development of corneal or conjunctival toxic effects as corneal epithelial defects or chronic conjunctival follicular reaction

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospital, Asyut, Egypt